CLINICAL TRIAL: NCT06281496
Title: AlloCare - Support and Management of Late Effects After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: AlloCare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Mette Schaufuss Engedal, Clinical nurse specialist, Ph.d student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Rigshospitalet, Hematology
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hematological Diseases
Keywords: Late effects. Survivorship. Allo-HSCT
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Intervention Model Description: One site, two arm randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention is a stepped-care multi-modal intervention and consists of 4 steps, including screening for vulnerability, digital health support and education. Individual consultations based on PRO data (HM-PRO) and multidisciplinary late effects management based on PRO assessment. The multidisciplinary team will consist of nurses, hematologists, physiotherapists, social workers, and dietitians.
  Interventions: Behavioral: AlloCare
- Control Group (No Intervention): Patients in the control group will receive usual care

INTERVENTIONS:
Behavioral: AlloCare — Survivorship supportive care
  Arms: Intervention group

SUMMARY:
A developed multimodal intervention targeting late effects in survivors of allogeneic hematopoietic stem cell transplantation (allo-HSCT) will be evaluated in a two-arm randomized controlled trial with an internal pilot phase.

DETAILED DESCRIPTION:
The study aims to investigate the effect of a stepped care intervention in allo-HSCT survivors on health-related quality of life and late effects.

Method:

This study is designed as a one-site, two-arm prospective randomized controlled trial proceeding an internal pilot phase.

Population/recruitment:

Recruitment, inclusion, and exclusion criteria as described in the eligibility section. Included patients will be randomized and allocated 1:1 to an intervention group or a control group.

Intervention:

a stepped-care multi-modal intervention

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age> 18 years) treated with myeloablative or non-myeloablative HSCT in outpatient follow-up without recurrent disease are eligible for inclusion.

Exclusion Criteria:

* Patients with recurrence or subsequent malignancy requiring cancer treatment or lack of access to email and the Internet will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life - summary score measured by European Organisation for Research and Treatment of Cancer QOL questionnaire (EORTC-QOL-C30) | 15 months (baseline 3, post intervention 12 and follow-up 18 month after treatment with allogeneic stem cell transplantation)
  Between-group changes in Quality of life - from baseline 3 months post treatment with allogenenic stem cell transplantation to postintervention 12 months post treatment with allogeneic stem cell transplantation. EORTC Quality of Life core questionnaire (QLQ-C30). The EORTC QoL Core Questionnaire EORTC QLQ-C30 is a 30-item instrument designed to measure quality of life in all cancer patients. The questionnaire consists of five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and some single items assessing additional symptoms commonly reported by cancer patients

SECONDARY OUTCOMES:
Survivorship specific quality of life | 15 months (baseline 3, post intervention 12 and follow up 18 month after treatment with allogeneic stem cell transplantation)
  EORTC-QOL-SURV100, Quality of life questionnaire applicable to cancerfree survivors. It consists of 100 questions divided over thirteen functional scales (i.e. Physical; Role ; Emotional; and Cognitive functioning; Body image; Symptom awareness; Positive health behavior change; Positive life outlook; Positive impact on behavior towards others; Positive social functioning; Work; Sexual functioning; Global health status), nine symptom scales (i.e. Social isolation; Fatigue; Pain; Sleep problems; Health distress; Negative health outlook; Social interference; Sexual problems), one Symptom checklist assessing chronic side effects of cancer treatments, and twelve single items.
  Score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QL represents a high QL, but a high score for a symptom item represents a high level of symptomatology.
Health literacy | 15 months (baseline 3, post intervention 12 and follow up 18 month after treatment with allogeneic stem cell transplantation)
  The survey encompasses nine separate scales exploring 9 different domains of health literacy. The following health literacy domains have been chosen; Scale 1: Feeling understood and supported by health care providers. Scale 3: Actively managing my health. Scale 8: Ability to find good health information and finally Scale 9: Understanding health information well enough to know what to do. The scales can be used individually as no summary score of total health literacy can be measured.
Referrals to municipality rehabilitation | 15 months (baseline 3, post intervention 12 and follow up 18 month after treatment with allogeneic stem cell transplantation)
  Municipal rehabilitation adresses both physical rehabilitation as well as psychosocial and work related problems based on disease and cancer treatment.
Modified 7-day Lee Chronic-versus-Host Disease Symptom Scale | 15 months (baseline 3, post intervention 12 and follow up 18 month after treatment with allogeneic stem cell transplantation)
  Validated questionnaire to measure degree of Graft Versus Host disease. The scale contains 28 items grouped in 7 subscales (skin, eye, mouth, lung, nutrition, energy, and psychological), and a 7 day recall period. Patients report how "bothered" they feel about each symptom over the previous 7 days using a five-point Likert scale from "not at all" to "extremely". range from 0 to 100, with a higher score indicating worse symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Mette Schaufuss Engedal, MSc, Principal Investigator — Rigshospitalet. Department of Hematology. Denmark; Mary Jarden, Study Director — Rigshospitalet. Department of Hematology. Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No